CLINICAL TRIAL: NCT04929795
Title: Effects of Music Beat on Motor Function in Individuals At Risk for Psychotic Onset and Schizophrenia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr WANG Shumei (Other)
Responsible Party: Sponsor-Investigator, Dr WANG Shumei, Assistant Professor, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20210610001
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Psychosis; Parkinsonism; Dyskinesias
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Parkinsonian Disorders; Dyskinesias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- at risk- RAS (Experimental): At-risk individuals in the experimental group will undergo upper-limb movement training with the aid of music beat serving as a type of rhythmic auditory stimulation (RAS).
  Interventions: Behavioral: Rhythmic auditory stimulation (RAS)
- at risk- no RAS (Active Comparator): At-risk individuals in the control group will receive upper-limb training without the aid of RAS.
  Interventions: Behavioral: no RAS
- schizophrenia- RAS (Experimental): Schizophrenia patients in the experimental group will undergo upper-limb movement training with the aid of RAS.
  Interventions: Behavioral: Rhythmic auditory stimulation (RAS)
- schizophrenia- no RAS (Active Comparator): Schizophrenia patients in the control group will receive upper-limb training without the aid of RAS.
  Interventions: Behavioral: no RAS

INTERVENTIONS:
Behavioral: Rhythmic auditory stimulation (RAS) — The song named 'Sign of The Times' is played and recorded by the research personnel beforehand. The beat of the song will serve as RAS. The computer software "Audacity" will be used to adjust tempi of RAS. Before intervention, the participant is required to execute the movement task without the aid of RAS as quickly as possible for 30 seconds, so that we obtain his/her baseline movement tempo. For each 40-minute training session in the first training week, three RAS tempi will be provided for the first, second, and last 10 minutes with a five-minute break in between: normal (100% of the baseline tempo), quick (105% of the baseline tempo), and fast (110% of the baseline tempo). With each training week, the three RAS tempi will be increased by 5%. Participants in the experimental groups are required to use their right hand to pick up beads from source bowls to the target bowl when listening to the song. The 3-week intervention program will include 21 40-minute daily training sessions.
  Arms: at risk- RAS; schizophrenia- RAS
Behavioral: no RAS — The training protocol will be the same as that used in the experimental group except the lack of RAS during execution of the movement task.
  Arms: at risk- no RAS; schizophrenia- no RAS

SUMMARY:
The purpose of this project is to investigate whether a 3-week training program involving music beat (serving as a type of rhythmic auditory stimulation) reduces the severity of bradykinesia and dyskinesia in at-risk individuals and schizophrenia patients. It is hypothesized that the program is effective in reducing the severity of bradykinesia and dyskinesia in at-risk individuals and schizophrenia patients.

ELIGIBILITY:
For at-risk participants:

Inclusion criteria:

1. A score of or above 9 in the Chinese version of the 16-item Prodromal Questionnaire (CPQ-16), or a score of or above 8.18 in the Chinese version of Community Assessment of Psychic Experiences with 15 items (CAPE-C15), or a score of or above 17 in Schizotypal Personality Questionnaire-Brief (SPQ-B);
2. an age of 13 years or above;
3. score > 60 in The Chinese version of Edinburgh Handedness Inventory (CH-EBI) to ensure right handedness; and
4. score ≥ 22 in Montreal Cognitive Assessment Hong Kong Version (HK-MoCA) to ensure no serious cognitive deficits so that they can understand instructions.

Exclusion criteria:

1. psychiatric diagnosis by self-report;
2. cardiovascular, neurological, muscular or orthopedic diseases that may affect hand movements;
3. taking psychiatric medications;
4. substance abuse; and
5. being pregnant.

For schizophrenia participants:

Inclusion criteria:

1. a diagnosis of schizophrenia without other psychiatric diseases;
2. the age ≥ 18 years;
3. score > 60 in CH-EBI to ensure right handedness; and
4. score ≥ 22 in HK-MoCA to ensure no serious cognitive deficits so that they can understand instructions.

Exclusion criteria:

1. cardiovascular, neurological, muscular or orthopedic diseases that may affect hand movements;
2. substance abuse; and
3. being pregnant.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right before the 1st session of the intervention
  normalized movement time (representing severity of bradykinesia). Unit: second/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right after the last session of the intervention
  normalized movement time (representing severity of bradykinesia). Unit: second/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right before the 1st session of the intervention
  normalized number of movement units (representing severity of dyskinesia). Unit: units/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right after the last session of the intervention
  normalized number of movement units (representing severity of dyskinesia). Unit: units/mm

CONTACTS AND LOCATIONS:
Locations (1):
- ST814, the Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang SM, Chan HY, Chan CY, Fong LY, Chan WL, Wu KY, Yip LC, Wong WY, Ng CL, Fong KNK. Effects of Music Rhythm on Movement Abnormalities in People With Psychotic-Like Experiences: A Pilot Randomised Controlled Trial Using Motion Analysis. Early Interv Psychiatry. 2025 Nov;19(11):e70111. doi: 10.1111/eip.70111. PMID 41254481